CLINICAL TRIAL: NCT05234541
Title: To Investigate the Value of the Cut-off Perfusion Index Showing That the Block is Successful in Infraclavicular Blocks Performed Under Ultrasound Guidance.
Brief Title: Measurement of Cut-off Perfusion Index Value in Infraclavicular Blocks
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, MEHMET DURAN, assistant professor, Adiyaman University
Other Study IDs: 2020/6-18; ISEYHANLI (Other: AdiyamanU)
Record Dates: First submitted 2022-02-01; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-07

CONDITIONS: Upper Extremity Surgery
Keywords: infraclavicular block, perfusion index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the value of the cut-off perfusion index showing that the block is successful in infraclavicular blocks performed under ultrasound guidance.

DETAILED DESCRIPTION:
In upper extremity procedures, ultrasound (US) guided infraclavicular block is a frequently used approach. Today, the frequency of studies on the perfusion index (PI), which can be used as a criterion in the evaluation of block success, is increasing. The aim of this study is to evaluate the success and effectiveness of infraclavicular approach block with perfusion index using ROC (Receiver Operating Characteristic) curves.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 PATIENTS
* PATIENTS BETWEEN 18-65 YEARS
* PATIENTS WITH INFRACLAVICULAR BLOCK

Exclusion Criteria:

* ASA3-4 PATIENTS
* PATIENTS UNDER THE AGE OF 18, PATIENTS OVER 65
* PATIENTS WHO DO NOT WANT TO BE INCLUDED IN THE STUDY
* PATIENTS WITH CONTRAINDICATION TO INFRACLAVICULAR BLOCK
* PATIENTS WITHOUT COOPERATION
* PATIENTS WITH DIABETES MELLITUS
* THOSE WHO HAVE PERIPHERAL ARTERY DISEASE

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA1-2 50 PATIENTS BETWEEN 18-65 YEARS
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
To Investigate the Value of the Cut-off Perfusion Index Showing That the Block is Successful in Infraclavicular Blocks Performed Under Ultrasound Guidance | Perfusion index, pulse and blood pressure will be measured 5-10-20 minutes after the block is made.
  To measure perfusion index values in patients aged 18-65 years who underwent upper extremity surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University Recruitment, Adıyaman, Turkey (Türkiye)